CLINICAL TRIAL: NCT06021509
Title: A Prospective, Multicenter, Single-arm Clinical Study of NovoClasp Transcatheter Mitral Valve Clip and Steerable Guide Catheter for Treating Moderate to Severe and Severe Degenerative Mitral Regurgitation (DMR)
Brief Title: Clinical Study of NovoClasp for Treating Moderate to Severe and Severe Degenerative Mitral Regurgitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Enlight Medical Technologies (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YM-2022-001
Record Dates: First submitted 2023-08-15; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Degenerative Mitral Valve Disease
Keywords: transcatheter edge-to-edge repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NovoClasp system (Experimental)
  Interventions: Device: NovoClasp® transcatheter mitral valve clip and steerable guide catheter

INTERVENTIONS:
Device: NovoClasp® transcatheter mitral valve clip and steerable guide catheter — The experimental device is a class III implanted valve device, which will be used to treat the mitral valve regurgitation via transcatheter edge-to-edge repair.
  Other Names: transcatheter edge-to-edge repair for mitral valve

SUMMARY:
To validate the safety and efficacy of transcatheter edge-to-edge repair (TEER) using the NovoClasp® transcatheter mitral valve clip and steerable guide catheter in the treatment of moderate to severe and severe degenerative mitral regurgitation (DMR).

DETAILED DESCRIPTION:
This trial is a prospective multi-center single-arm confirmatory study. A total of 102 subjects will be enrolled in multiple centers nationwide. Subjects who meet the trial requirements, fulfill the inclusion criteria, voluntarily participate in the study, and provide informed consent will undergo mitral edge-to-edge repair using the NovoClasp® transcatheter mitral valve clip system and steerable guide catheter for the treatment of moderate to severe or severe degenerative mitral regurgitation (DMR). Follow-up assessments will be conducted at discharge, as well as at 30 days, 90 days, 180 days, and 360 days postoperatively. The primary endpoint will be the treatment effectiveness rate at 360 days post-surgery. Secondary endpoint measures include treatment effectiveness at other time points, surgical success rate, all-cause mortality, device/procedure-related mortality, incidence of adverse events, and serious adverse event rates. The trial aims to comprehensively assess the safety and efficacy of the NovoClasp® transcatheter mitral valve clip and steerable guide catheter produced by Enlight Medical Technologies (Shanghai) Co., Ltd..

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for this study.

1. Age 18 years.
2. Willingness to comply with the protocol requirements and data collection procedures, ability to understand the purpose of the trial, voluntary participation, and signing of informed consent by the subject or legal guardian.
3. Confirmation by echocardiography of moderate to severe (3+) or severe (4+) degenerative mitral regurgitation.
4. Echocardiography showing left ventricular ejection fraction 30%, left ventricular end-systolic diameter (LVESD) 60mm, and pulmonary artery systolic pressure (PASP) 70 mmHg.
5. NYHA functional classification II-IV.
6. Presence of a primary regurgitant jet; if a secondary regurgitant jet is present, it should be clinically insignificant based on investigator assessment.
7. Evaluated by a multidisciplinary team as suitable for the investigational procedure using the study device.
8. Society of Thoracic Surgeons (STS) score 4 or evaluated as high surgical risk for mitral valve repair by two cardiac surgeons.

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for this study.

1. History of prior mitral valve surgery or heart transplant.
2. Severe organ dysfunction that may affect study evaluation, including but not limited to:

   1. Right heart failure or biventricular heart failure.
   2. Severe restrictive or obstructive lung disease (COPD) requiring continuous oxygen therapy or oral steroid treatment.
   3. Severe renal insufficiency requiring or likely to require continuous renal replacement therapy (CRRT) or dialysis postoperatively.
   4. Severe carotid artery stenosis confirmed by imaging to be >70%.
3. History of cerebrovascular accident within the past 1 month.
4. Acute deep vein thrombosis or acute pulmonary embolism history.
5. Any known active infection.
6. Active infective endocarditis (eligible 6 weeks after standard antimicrobial treatment), rheumatic heart valve disease, or radiation-induced valve disease.
7. Cardiac or major vascular surgical or interventional procedure within 30 days (coronary angiography is allowed).
8. Coexisting moderate or greater valvular disease (aortic valve, tricuspid valve, pulmonary valve stenosis or regurgitation).
9. Known other cardiac or major vascular diseases requiring surgical or interventional intervention, including but not limited to coronary artery disease, myocardial disease, aortic disease (except for coronary angiography).
10. Echocardiographic evidence of intracardiac mass, thrombus, vegetation, or mitral valve orifice area (MVOA) 4.0 cm2, or any condition unsuitable for the study device, including but not limited to:

    1. Unsuitable for leaflet capture due to severe calcification or cleft.
    2. Lack of primary and secondary chordal support in the capture area.
    3. Leaflet free edge length < 0.8 cm.
11. Known conditions that preclude study procedure (including but not limited to allergies to device components, coagulation disorders, life expectancy < 1 year).
12. Pregnant or breastfeeding women or those planning pregnancy during the trial period.
13. Intending or currently participating in another interventional clinical trial.
14. Other conditions deemed inappropriate for participation in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-06-25 (Estimated); Study Completion 2028-06-25 (Estimated)

PRIMARY OUTCOMES:
Treatment effectiveness rate | 1 year
  Treatment effectiveness is defined as the success of the procedure with the mitral valve regurgitation sustained at moderate or lower (<=2+) after the surgery, without major adverse events or secondary interventions (interventional or surgical).

SECONDARY OUTCOMES:
Procedural success rate | immediately after procedure
  Successful implantation of a single device as intended by the operator, successful retrieval of the delivery system, absence of device migration, dislodgment, embolization, related complications, or other unforeseen incidents.
Procedural success rate | During the perioperative period
  Defined as successful completion of the investigational procedure as intended by the operator (implantation of at least 1 study device) and reduction of mitral valve regurgitation to moderate or below (<=2+), without open surgery, major adverse events during the perioperative period, or secondary interventions (interventional or surgical).
  Note: Major adverse events include cardiovascular-related deaths, stroke, myocardial infarction, need for renal replacement therapy, severe bleeding (hemoglobin decrease >=3g/dL compared to baseline, or requiring >=3 units of blood transfusion), or organ damage, failure, or death dur to blood loss.
Rate of Treatment success | 30 days, 180 days
  Treatment effectiveness is defined as the success of the procedure with the mitral valve regurgitation sustained at moderate or lower (<=2+) after the surgery, without major adverse events or secondary interventions (interventional or surgical).
Changes in New York Heart Association (NYHA) Functional Classification | through study completiong, an average of 1 year.
  The NYHA Classification provides nomenclature to describe an overall cardiac appraisal of the status of a patient with heart disease.
  Class I: Patients with cardiac disease but without resulting limitation of physical activity.
  Class II: patients with cardiac disease resulting in slight limitation of physical activity.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Patient with cardiac disease resulting in inability to carry on any physical activity without discomfor.

OTHER OUTCOMES:
All cause mortality | through study completion, an average of 1 year
Device/Procedure-related mortality | through study completion, an average of 1 year
Major adverse events | through study completion, an average of 1 year
Serious adverse events | through study completion, an average of 1 year
Number of participants with device-related adverse events | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China